CLINICAL TRIAL: NCT03451981
Title: Evaluation of the Adjunctive Use of Er:YAG Laser or Erythritol Air-polishing in the Non-surgical Treatment of Peri-implantitis: a RCT
Brief Title: Non Surgical Protocol for Treatment of Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Clementini, Principal Investigator, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: peri-implant non surgical-1
Record Dates: First submitted 2018-02-20; First posted 2018-03-02 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Peri-Implantitis
Keywords: non surgical therapy; laser; air powder
MeSH Terms: conditions — Peri-Implantitis | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mechanical instrumentation with curettes (Sham Comparator): mechanical instrumentation: Inflammatory tissue, excess cement or plaque deposits will be removed using hand instruments (titanium curettes) and the implant surface will be cleaned.
  Interventions: Procedure: mechanical instrumentation
- Er:YAG laser (Experimental): Er:YAG laser treatment will be provided on the implant surface.
  Interventions: Procedure: mechanical instrumentation; Procedure: Er:YAG laser
- Air Powder (Active Comparator): an Air-Powder treatment will be provided on the implant surface.
  Interventions: Procedure: mechanical instrumentation; Procedure: Air Powder

INTERVENTIONS:
Procedure: mechanical instrumentation — mechanical debridement: Inflammatory tissue, excess cement or plaque deposits will be removed using hand instruments (titanium curettes) and the implant surface will be cleaned
  Other Names: titanium curettes
Procedure: Er:YAG laser — mechanical debridement: Inflammatory tissue, excess cement or plaque deposits will be removed using hand instruments (titanium curettes) and the implant surface will be cleaned. Furthermore, Er:YAG laser treatment will be provided on the implant surface.
  Arms: Er:YAG laser
Procedure: Air Powder — mechanical debridement: Inflammatory tissue, excess cement or plaque deposits will be removed using hand instruments (titanium curettes) and the implant surface will be cleaned. Furthermore, an Air-Powder treatment will be provided on the implant surface.
  Arms: Air Powder

SUMMARY:
Peri-implantitis is an important disease entity as a result of its high prevalence and the lack of a standard mode of therapy.

Non-surgical therapy of peri-implant disease, especially when bone loss is not high, appears to be partially effective in resolving the disease. In several cases, however, only limited improvements have been reported in the main clinical parameters (bleeding at the survey and presence of the pocket) and there is a clear tendency to relapse of the disease.

In these cases it is therefore recommended to consider adjunctive therapies. Numerous approaches have been used for implant surface decontamination including mechanical, chemical and treatments by means of air-powder or laser.

The aim of the present randomized controlled clinical trial will be to assess the efficacy in improving clinical parameters of two further methods of implant surface decontamination (Er:YAG laser or air-abrasive device) after mechanical cleaning during non surgical treatment of peri-implantitis.

DETAILED DESCRIPTION:
Peri-implantitis, defined as an inflammatory lesion in the surrounding peri-implant tissues with loss of supporting bone, is an important disease entity as a result of its high prevalence and the lack of a standard mode of therapy. Although the current epidemiological data are limited, peri-implantitis affects 28-56% of the subjects and 12-43% of the implants.

Numerous approaches have been used for implant surface decontamination during peri-implant surgery, including mechanical, chemical and laser treatments. Using conventional mechanical means, eradication of pathogens on implant surfaces with threads and often with rough surface structures is difficult. Treatment models, such as debridment, effectively used to treat teeth with periodontitis, cannot be used in the same way on rough threaded implant surfaces. The implant rough surface structure also provides the bacteria with ''protected areas'', inaccessible to conventional mechanical removal.

A treatment protocol that may offer an advantage over traditional mechanical treatment includes the use of laser therapy. Data have shown that treatments with Er:YAG lasers have a bactericidal effect. Er:YAG laser treatment can debride the implant surface effectively and safely. Slightly better clinical results in terms of bleeding on probing and clinical attachment level have been reported by Er:YAG laser treatment as compared with traditional non-surgical mechanical debridement with curette and chlorhexidine.

The air abrasive method for the removal of bacterial plaque on tooth surfaces has also been used in the treatment of peri-implantitis, demonstrating no relevant adverse effects. Until recently, air-polishing devices have used a slurry of water and sodium bicarbonate (NaHCO3) and pressurized air/water. A less abrasive method using an amino acid glycine has been proven to be effective in removing bacterial biofilm structures in deep periodontal pockets and safe by not causing emphysema. Moreover the use of a glycine-based powder does not seem to cause titanium implant surface changes.

The aim of the present randomized controlled clinical trial will be to assess the efficacy in improving clinical parameters of two further methods of implant surface decontamination (Er:YAG laser or air-abrasive device) after mechanical cleaning during non surgical treatment of peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least one screw-type titanium implant exhibiting bleeding and/or suppuration on probing combined with:

  1. a PPD ≥ 5 mm and bone loss > 2 mm (compared to crestal bone levels at the time of placement of the reconstruction)
  2. a PPD ≥ 6 mm and bone loss ≥ 3 mm (not compared to crestal bone levels at the time of placement of the reconstruction)
* single tooth and bridgework restorations without overhangings
* no evidence of occlusal overload (i.e. occlusal contacts revealed appropriate adjustment)
* implant function time ≥ 1 year.

Exclusion Criteria:

* Patients with uncontrolled diabetes,
* patients with osteoporosis or under bisphosphonate medication,
* pregnant or lactating women,
* patients with a history of radiotherapy to the head and neck region
* patients with incapability to perform basal oral hygiene measures due to physical or mental disorders
* hollow implants
* implant mobility
* implants at which no position could be identified where proper probing measurements could be performed;
* previous surgical treatment of the peri-implantitis lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
probing pocket depth changes | baseline, 1, 3, 6 months
  changes in probing pocket depth, measured from the mucosal margin to the bottom of the pocket

SECONDARY OUTCOMES:
Bleeding on probing changes | baseline,1, 3, 6 months
  changes of bleeding on probing, evaluated as present if bleeding will be evident within 30 s after probing, or absent, if no bleeding will be noticed within 30 s after probing
endpoint of therapy | 1,3,6 months
  residual PPD ≤5 mm with BoP present at no more than one site and no SoP (Tonetti et al., 2023), assessed at the implant level.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo De Sanctis, Prof., Study Chair — University Vita Salute San Raffaele
Locations (1):
- Università Vita-Salute San Raffaele, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided